CLINICAL TRIAL: NCT03170492
Title: Does Computerized Cognitive Training Improve Executive Functioning in the Older Adult?
Acronym: CCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Sciences in Philadelphia (Other)
Collaborators: GenesisCAREs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 947324
Record Dates: First submitted 2017-05-22; First posted 2017-05-31 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Cognitive Impairment, Mild; Executive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Training (Experimental): RehaCom for 480 minutes over 12 weeks.
  Interventions: Other: RehaCom Computerized Cognitive Training for 480 minutes
- Pencil-and-Paper Cognitive Training (Active Comparator): Table-top based activities for 480 minutes over 12 weeks.
  Interventions: Other: Pencil-and-Paper Cognitive Training for 480 minutes

INTERVENTIONS:
Other: RehaCom Computerized Cognitive Training for 480 minutes — Student OT doctoral researchers will guide the subject when participating in the RehaCom program. RehaCom is computer hardware and software designed for assisted cognitive rehabilitation. The program is designed to target specific aspects of attention, concentration, memory, perception, and problem-solving. As the training goes on, the tasks will become easier or harder depending on the subject's performance. The first session will begin with a screening module with an example and a practice session to make sure the client understands the task. After screening, the results page shows the subject's performance compared with age-matched norms. This gives a helpful indication as to the severity of the deficit and advises the researcher on the particular training module to be used. The subject will continue the training modules for a total of 480 minutes of training over 12 weeks.
  Arms: Computerized Cognitive Training
Other: Pencil-and-Paper Cognitive Training for 480 minutes — Student OT doctoral researchers will engage the subject in various pen-and-paper exercises designed to improve cognitive functions: attention and concentration, memory, language, calculation, and orientation. These could include, but are not limited to: word puzzles, calculation or number puzzles, and map reading. The subject will continue the training modules for a total of 480 minutes of training over 12 weeks.
  Arms: Pencil-and-Paper Cognitive Training

SUMMARY:
Explanation of the study: As the older adult population continues to rise, so will normal cognitive aging. This increase raises concern for maintaining cognitive function and possibly delaying the onset of disorders such as dementia. Cognitive training (CT) is one potential solution which may be done using computer programs, pencil-and-paper problem solving activities, or everyday tasks. Traditional, skilled occupational therapy (OT) is not reimbursed for this type of preventative or maintenance services. CT may be a fundable answer for older adults to maintain or even improve cognitive function. The purpose is to determine if computerized CT, utilizing a specific program (RehaCom), improves executive functioning in the older adult with mild cognitive impairment, as compared to pencil-and-paper CT.

How study is performed: Participants who meet the inclusion criteria will complete a 9-question demographic survey and pre-test standardized cognitive tests. The experimental group will complete RehaCom computer training and the control group will complete paper-and-pencil based training. All trainings will take place at Mercy LIFE and will be conducted by trained OT students. Subjects will complete a total of 480 minutes of training over a 12-week period, within 30 to 60 minutes sessions. After the 480 minutes of training, subjects will complete the cognitive post-tests.

How data is collected, de-identified and analyzed: Participants who enroll will be assigned a code number linked to their first and last name. This coding will de-identify participants before analyzing or reporting. All signed forms, data collected, and data identified will be kept in a locked cabinet in the researcher's office. All stored files will be shredded one year after the study.

Interventions/tests/medications:

Computerized CT: RehaCom is a computer program that was designed to assist cognitive rehabilitation. The program targets attention, concentration, memory, perception, and problem-solving, with trainings lasting for a total of 480 minutes over 12 weeks.

Pencil-and-paper CT: Various pencil-and-paper exercises to improve attention, concentration, memory, language, and orientation will be used. Such exercises may include word puzzles, calculation or number puzzles, and map reading, for a total of 480 minutes of training over 12 weeks.

Potential risks: Risks of feeling segregated are minimal, as all members have been offered the opportunity to use the site's computer room. Risks may include cognitive fatigue (in both groups) or overstimulation during computer use. Breaks will be given at any sign of these symptoms. There is a small possibility that the participant may become too overwhelmed or stressed with the cognitive training. Upon notice of these symptoms, activities will cease immediately.

Potential and expected benefits: Participants may gain a greater insight into cognitive abilities and improvement of executive functioning skills. Increased knowledge on effects of using cognitive software in a community-based setting may also occur. Mercy LIFE will receive the benefit of continued use of the RehaCom software and laptop as the equipment will be left at the site. Additionally, these findings may help other community-based sites incorporate specific cognitive training for other older adults.

DETAILED DESCRIPTION:
As baby boomers age, physical engagement recommendations are well known, but the issue of maintaining cognitive function continues to be problematic. Researchers have suggested that individuals who are engaged in intellectual activities in middle and late adulthood fare better cognitively than their less engaged peers (Singh-Manoux, Richards, & Marmot, 2003). Research has shown that playing videogames can improve several aspects of cognition, including fluid general intelligence (Jaegii, Buschkuel, Jonides, & Shah, 2011) and attentional and perceptual functioning (Green & Bavelier, 2007). Gaitán et al. (2013) reported that when computer-based cognitive training was provided as an adjunct to pen-and-paper training for individuals with mild cognitive impairment, positive influences in memory and decision-making were observable. In regards to computer-based training for the healthy community-dwelling older adult to prevent cognitive decline, this evidence is becoming more promising. In the "ACTIVE" study, one of the largest, longest-term studies to date, 2,785 participants were randomized to four groups, with only the computerized speed training group showing a statistically significant impact on preventing cognitive decline. At ten years, the researchers observed a 33 percent reduction in risk of developing dementia over the time of the study (Alzheimer's Association, 2016; Rebok et al., 2014). Traditional, skilled occupational therapy is not reimbursed for these types of preventative, maintenance-type services. As the aging population continues to rise, so will the incidence of normal cognitive aging. Community or home-based cognitive training may be a fundable answer for older adults to maintain or even improve cognitive function.

Considering the older adult with known mild cognitive impairment, this evidence is emerging. The current consensus is that there is a lack of significant evidence to support the use of computer-based cognitive training alone and the recommendation is to obtain "real-world" measurements of the transfer to everyday skills (Muller, 2016). The investigators will utilize the Executive Function Performance Test (EFPT) to gain a reliable depiction of the participant's current executive function as it relates to performance of daily tasks. Both skill-based and performance-based measures will be used throughout the study to capture various areas of the participants' cognition. The investegators will focus the study on computerized cognitive training utilizing a specific program (RehaCom) in a single community-based setting to address the older adult's executive functioning.

Primary research question: Does computerized cognitive training improve skill-based executive functioning skills in the older adult, as compared to traditional cognitive training? Secondary research question: Does computerized cognitive training improve performance-based executive functioning skills in the older adult, as compared to traditional cognitive training?

The population for this project will be selected via convenience sampling from Mercy LIFE West Philadelphia. Please see "Eligibility Criteria" section for inclusion criteria.

Recruiting older adults that may live with cognitive impairment is necessary to investigate the possible positive effects for this growing population. Published evidence is emerging and ongoing for older adults without cognitive impairment, but researchers recommend the further investigation of the effect of cognitive training on individuals with mild cognitive impairment.

Subjects will be randomized to one of two groups: (1) computerized cognitive training or (2) pencil-and-paper traditional cognitive training.

Members of Mercy LIFE West Philadelphia are provided with transportation to the center for their normal activities. The members will participate in cognitive training sessions (computerized cognitive training vs. pencil-and-paper traditional cognitive training) 30-60 minutes per session, to total 480 minutes of training, within 12 weeks, at times that the participant has available throughout the day and week at the center. The researchers will keep a coded, detailed log of the session length to total the minutes completed throughout the 12 weeks. This flexibility of dosing (length, frequency, and duration) is at the request of Mercy LIFE West Philadelphia's Research Committee, to respect the members' medical and activity schedules.

Group 1 (computerized cognitive training): Student OT doctoral researchers will guide the subject when participating in the RehaCom program. RehaCom is computer hardware and software designed for assisted cognitive rehabilitation. The program is designed to target specific aspects of attention, concentration, memory, perception, and problem-solving. As the training goes on, the tasks will become easier or harder depending on the subject's performance. The first session will begin with a screening module with an example and a practice session to make sure the client understands the task. After screening, the results page shows the subject's performance compared with age-matched norms. This gives a helpful indication as to the severity of the deficit and advises the researcher on the particular training module to be used. The subject will continue the training modules for a total of 480 minutes of training over 12 weeks.

Group 2 (pencil-and-paper traditional cognitive training): Student OT doctoral researchers will engage the subject in various pen-and-paper exercises designed to improve cognitive functions: attention and concentration, memory, language, calculation, and orientation. These could include, but are not limited to: word puzzles, calculation or number puzzles, and map reading. The subject will continue the training modules for a total of 480 minutes of training over 12 weeks.

All of the following will be administered by the researchers prior to the 480 minutes of training sessions, as well as upon completion after the 480 minutes of training to assess overall cognitive performance and executive functioning. Please see "Outcome Measures" section for details on the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Members of Mercy LIFE West Philadelphia
* 55 years of age and older
* Initial score of ≥20/30 on the Mini Mental State Examination (MMSE)
* A current score of ≥17/30 on the Montreal Cognitive Assessment (MoCA)
* Visual skills required to adequately view images on computer screens and paper, assessed by the subject's ability to read the information in the informed consent.

Exclusion Criteria:

* Younger than 55 years old
* MMSE score < 21/30
* MoCA <18
* Inability to visually read information in the informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-11-03 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 10 minutes
  Montreal Cognitive Assessment (MoCA): The MoCA was developed as a more challenging test that includes executive function, higher-level language, and complex visuospatial processing to enable detection of mild impairment with less ceiling effect than the MMSE.
Delis-Kaplan Executive Functioning System (Letter Fluency) | 5 minutes
  Delis-Kaplan Executive Functioning System (D-KEFS) Verbal Fluency Test: Measures letter fluency. The evaluator instructs the subject, "I'm going to say a letter of the alphabet. When I say begin, I want you to tell me as many words as you can that begin with that letter. You will have 60 seconds before I tell you to stop. None of the words can be names of people, or places, or numbers." Score is obtained as the number of words recalled (duplicates or errors removed).
Trail Making Test Part A | 3 minutes
  The Trail Making Test Part A: A test of visual conceptual and visuo-motor tracking. TMT-A measures attention, visual search and motor function; scored as time to completion.
Trail Making Test Part B | 4 minutes
  The Trail Making Test Part B: A test of visual conceptual and visuo-motor tracking. TMT-B measures executive functioning, speed of attention, visual search and motor function; scored as time to completion.

SECONDARY OUTCOMES:
Executive Function Performance Test | 30 minutes
  • Executive Function Performance Test (EFPT): The EFPT assesses the performance of four selected tasks that are essential for self-maintenance and independent living, such as oatmeal preparation, using the telephone, taking medication and paying bills. Each task has five items: initiation, organization, sequencing, judgment and safety, and completion, defined as executive functions. The total score is the sum of the performance on all four tasks, scored from 0 - 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Benham, OTD, Principal Investigator — University of the Sciences in Philadelphia
Locations (1):
- Mercy LIFE- West Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer's Association. (2016, July 27). New reports from the Alzheimer's Association International Conference® 2016. Retrieved from: https://www.alz.org/aaic/releases_2016/wed_300_ET.asp
- [Background] Baum, C. & Wolf, T. (2013). Executive Function Performance Test (EFPT). Retrieved from http://www.ot.wustl.edu/about/resources/executive-function-performance-test-efpt-308
- [Background] Delis, D.C., Kaplan, E. & Kramer, J.H. (2001). The Delis-Kaplan Executive Function System. San Antonio, TX: The Psychological Corporation.
- [Background] Green CS, Bavelier D. Action-video-game experience alters the spatial resolution of vision. Psychol Sci. 2007 Jan;18(1):88-94. doi: 10.1111/j.1467-9280.2007.01853.x. PMID 17362383
- [Background] Gaitan A, Garolera M, Cerulla N, Chico G, Rodriguez-Querol M, Canela-Soler J. Efficacy of an adjunctive computer-based cognitive training program in amnestic mild cognitive impairment and Alzheimer's disease: a single-blind, randomized clinical trial. Int J Geriatr Psychiatry. 2013 Jan;28(1):91-9. doi: 10.1002/gps.3794. Epub 2012 Apr 3. PMID 22473855
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Shah P. Short- and long-term benefits of cognitive training. Proc Natl Acad Sci U S A. 2011 Jun 21;108(25):10081-6. doi: 10.1073/pnas.1103228108. Epub 2011 Jun 13. PMID 21670271
- [Background] Muller, K. D. (2016). A review of computer-based cognitive training for individuals with mild cognitive impairment and Alzheimer's Disease. Perspectives of the ASHA Special Interest Groups, 1(2), 47-61.
- [Background] Mungas D. In-office mental status testing: a practical guide. Geriatrics. 1991 Jul;46(7):54-8, 63, 66. PMID 2060803
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] National Institute on Aging. (2014). Cognitive training shows staying power [Press Release]. Retrieved from https://www.nia.nih.gov/newsroom/2014/01/cognitive-training-shows-staying-power
- [Background] Rebok GW, Ball K, Guey LT, Jones RN, Kim HY, King JW, Marsiske M, Morris JN, Tennstedt SL, Unverzagt FW, Willis SL; ACTIVE Study Group. Ten-year effects of the advanced cognitive training for independent and vital elderly cognitive training trial on cognition and everyday functioning in older adults. J Am Geriatr Soc. 2014 Jan;62(1):16-24. doi: 10.1111/jgs.12607. Epub 2014 Jan 13. PMID 24417410
- [Background] Singh-Manoux A, Richards M, Marmot M. Leisure activities and cognitive function in middle age: evidence from the Whitehall II study. J Epidemiol Community Health. 2003 Nov;57(11):907-13. doi: 10.1136/jech.57.11.907. PMID 14600119
- [Background] Strauss, E., Sherman, E.M.S. & Spreen, O. (2006) Trail making test. In: A Compendium of Neuropsychological Tests. New York: Oxford University Press, 655-659.
- [Background] Trzepacz PT, Hochstetler H, Wang S, Walker B, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Relationship between the Montreal Cognitive Assessment and Mini-mental State Examination for assessment of mild cognitive impairment in older adults. BMC Geriatr. 2015 Sep 7;15:107. doi: 10.1186/s12877-015-0103-3. PMID 26346644